CLINICAL TRIAL: NCT07405008
Title: Effect of Laser Acupuncture on Carpal Tunnel Syndrome Post Aromatase Inhibitors in Breast Cancer Patient .
Brief Title: Laser Acupuncture on Carpal Tunnel Syndrome .
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Naiera Sabry Mohamed Shams, Physiotherapy Specialist at Damanhur Medical National Institute, EL-Behira, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1172027
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Carpal Tunnel Syndrome (CTS) in Breast Cancer Patients
Keywords: LASER ACUPUNCTURE -CARPAL TUNNEL SYNDROME -AROMATASE INHIBITORS-BREAST CANCER PATIENT
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LASER acupuncture technique plus traditional physical therapy (Experimental): Group A: 27 patients ,suffered from CTS post breast cancer treatment with Aromatase inhibitors, will receive Laser acupuncture technique in addition to traditional physical therapy program (myofascial release, nerve flossing ex., Tendon gliding ex. strengthening ex., ROM ex. and night splint)3 times per week for 8 weeks.
  Interventions: Device: LASER acupuncture technique
- Traditional physical therapy program (Experimental): Group (B): 27 patients ,suffered from CTS post breast cancer treatment with Aromatase inhibitors , will receive traditional physical therapy program (myofascial release, nerve flossing ex., Tendon gliding ex., strengthening ex., ROM ex. and night splint) 3 times per week for 8 weeks.
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Device: LASER acupuncture technique — LASER Acupuncture technique:
  * Device: PR999, Medical Italia, Italy.
  * Maximum frequency: 5000 Hz
  * Dosage: 4j/point
  * Wave length :830 nm
  * Power output :50 m.W
  * Duration:12 min.
  * Frequency of treatment: 3 sessions/week.
  * Total treatment period: 8 weeks.
  * Total number of sessions: 24 sessions. The laser device will be positioned perpendicular to the skin over CTS area especially over each acupuncture point, for one minute duration for each point and the sessions will be conducted three times a week for eight weeks .
  Arms: LASER acupuncture technique plus traditional physical therapy
Other: Traditional physical therapy — Active assisted ROM exercises. Each exercise was performed for all movements namely flexion, extension, ulnar & radial deviations, supination and pronation, one set of each 10-15 repetitions within pain-free range and instructed to carry out their ADLs, Patient education regarding work modification and ergonomic recommendations and Tendon gliding exercises. Each exercise begins with the wrist and fingers fully extended. During tendon-gliding exercises, the fingers were placed in five discrete positions: straight, hook, tabletop, full fist and straight fist .
  Arms: Traditional physical therapy program

SUMMARY:
The study will be carried out on a total number of fifty-four females with age ranged 40 - 60 years old suffering from CTS post mastectomy ,the patients will be randomly assigned into two groups equal in number (27 patients for each group from Damanhur Medical National institute).

1. -Group (A): This group will include 27 patients will receive laser acupuncture technique 3 times per week in addition to traditional physical therapy program (myofascial release, nerve flossing ex., Tendon gliding ex. strengthening ex., ROM ex. and night splint) for 8 weeks.
2. -Group (B): This group will include 27 patients will receive traditional physical therapy program (myofascial release, nerve flossing ex., Tendon gliding ex., strengthening ex., ROM ex. and night splint) for 8 weeks.

DETAILED DESCRIPTION:
The study will be carried out on a total number of fifty-four females with age ranged 40 - 60 years old suffering from CTS post mastectomy , the patients will be randomly assigned into two groups equal in number (27 patients for each group from Damanhur Medical National institute).

1. -Group (A): This group will include 27 patients will receive laser acupuncture technique 3 times per week in addition to traditional physical therapy program (myofascial release, nerve flossing ex., Tendon gliding ex. strengthening ex., ROM ex. and night splint) for 8 weeks.
2. -Group (B): This group will include 27 patients will receive traditional physical therapy program (myofascial release, nerve flossing ex., Tendon gliding ex., strengthening ex., ROM ex. and night splint) for 8 weeks.

Equipment:

1. Measurement equipment:

   1. Nerve Conduction Studies (NCSs)
   2. Boston Carpal Tunnel Questionnaire (BCTQ)
   3. Hand-Held Dynamometer
2. Therapeutic equipment:

   1. Laser Acupuncture technique for group (A).
   2. Traditional Physical therapy program for both groups.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:

  * Patients' age will be ranged between 40-60 years old.
  * 54 Female patients had breast cancer will participate in this study.
  * All patients will have wrist pain and disability post AIS.
  * All patients will suffer from moderate to severe pain.
  * All patients will enroll to the study will have their informed consent

Exclusion Criteria:

* The potential participants will be excluded if they met one of the following criteria:

  * Patients with previous history of fracture at the wrist fracture.
  * History of any arthritis related to wrist.
  * Rheumatoid arthritis wrist secondary to fracture, dislocation,
  * Reflex sympathetic dystrophy and neurological disorder, Malignancy.
  * Epilepsy or any psychological disorders.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 54 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Median Motor Nerve Conduction Study | 8weeks
  With the help of electrode /conducting jelly, the recording was placed closed to motor of Abductor Policis Brevis and referance electrode 3 cm distal at the metacarpophalangeal joint. The ground electrode is placed between stimulation and recording electrode. A supramaximal stimulation was given at first to wrist and then at below. The difference between two latent period in msec gives the time taken by the impulses to travel from the elbow to the wrist.
Median Sensory Nerve Conduction Study: | 8 weeks
  The Orthodromic conduction recording was done in this case. Here the recording electrode was placed 3cm proximal to the distal wrist crease 3cm proximal to the recording electrode. The ring electrode were placed in the second and third digit and it was used for stimulation of the nerve with the cathode placed at the proximal inter phalangeal. The grounding electrode was placed between stimulating electrode and grounding electrode.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire (BCTQ) | 8weeks
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a widely recommended patient-reported outcome measure to evaluate symptoms and functions in carpal tunnel syndrome (CTS) patients. The BCTQ is a disease-specific PROM for CTS patients. It contains 2 measurement scales: a symptom severity scale (BCTQ-S) and a functional status scale (BCTQ-F). The BCTQ-S uses 11 questions to evaluate the intensity and frequency of pain, numbness, weakness and loss of dexterity on a five-point scale ranging from 1 (no symptoms) to 5 (severe symptoms). The results are interpreted as the average scores of the 11 questions. The BCTQ-F has 8 questions to evaluate the level of difficulty in performing daily tasks, each rated on a five-point scale ranging from 1 (no diffculty) to 5 (cannot do at all due to hand or wrist symptoms). The results are interpreted as the average scores of the 8 questions
Hand-Held Dynamometer (HHD) | 8weeks
  Hand-held dynamometers are portable devices usually incorporating a wireless load cell with an inbuilt microprocessor to measure isometric muscle force with good to excellent reliability across both clinical and healthy populations. These characteristics have made hand-held dynamometers a feasible and widely used tool to quantify muscle strength in a range of clinical populations. To assess hand grip, participants were seated comfortably in a chair with their feet supported. The hand and forearm being assessed was positioned with the shoulder adducted and in neutral rotation, with the elbow in 90◦ of flexion, forearm in neutral, and the wrist in 0 to 30◦ of extension and 0 to 15◦ of ulnar deviation. The participant was asked to grasp the hand-held dynamometer with the fingers wrapped around the handle. The clinical evaluator instructed the participant to perform a maximal contraction lasting three to five seconds, saying, "when I say go, I want you to squeeze the handle as hard as you

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethical Committee Faculty of Physical Therapy, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt